CLINICAL TRIAL: NCT06875778
Title: Development and Validation of Pregnancy Specific Pelvic Floor Rehab Protocol
Brief Title: Development & Validation of Pregnancy Specific Pelvic Floor Rehab Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sanna
Record Dates: First submitted 2025-02-20; First posted 2025-03-13 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Pelvic Floor Disorder; Pelvic Floor Muscle Weakness; Pelvic Floor Muscle Training; Pregnancy
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Intervention Model Description: This will be a Pretest- Post test Study Design with assignment of Patients in 1 group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pelvic Floor Rehab Group (Experimental): This Group will receive a developed Pelvic floor exercises protocol for 4 Weeks
  Interventions: Other: Pelvic Floor Exercises

INTERVENTIONS:
Other: Pelvic Floor Exercises — Low intensity Warm Up Pelvic Floor Exercises and Cool down training

SUMMARY:
Pelvic Floor Weakness is very common Facing by women during Pregnancy. PFM weakness is recognized as one of the problems encountered in patients with urinary and fecal incontinence which have very negative impact on Quality of life of Patients. This project aims to design, implement, and validate a pelvic floor rehabilitation protocol specifically for pregnant individuals.

DETAILED DESCRIPTION:
The review of existing literature undergoes the critical need for a pregnancy-specific pelvic floor rehab protocol to address the unique physiological and functional changes experienced during and after pregnancy. While current pelvic floor rehab approaches provide valuable insights, they often lack specific adaptations for the pregnant population, In First Phase of Study the protocol will be developed .The protocol will focus on preventing and managing pelvic floor dysfunction (PFD), such as urinary incontinence, pelvic organ prolapse, and pelvic pain, which are common during pregnancy. The program will incorporate evidence-based exercises, education, and lifestyle modifications, ensuring it is safe, effective, and adaptable to pregnancy.

In Second Phase it will be validated and Pilot testing will be done.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed pelvic floor dysfunction. Female participants experience pelvic floor symptoms such as incontinence, pelvic pain, or prolapse.

No previous participation in a structured pelvic floor rehabilitation program within the last six months

Exclusion Criteria:

* Pregnant women or those planning to become pregnant during the study period.
* Patients with neurological disorders affecting pelvic floor function (e.g., multiple sclerosis, spinal cord injury).
* Individuals with severe psychiatric conditions that might interfere with participation.
* Recent pelvic surgery within the last three months.
* Any contraindications to physical therapy or specific exercises included in the rehab program.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Gender must be Female
Enrollment: 15 (Actual)
Dates: Start 2024-02-11 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Pelvic Floor Distress Inventory (PFDI) | Baseline to 4th Week
  The PFDI-20 questionnaire is designed to evaluate symptoms and quality of life relating to PFDs; it has 20 items and three scales for three different symptoms to assess symptoms of distress from UI (Urinary Distress Inventory-6), POP (Pelvic Organ Prolapse Distress Inventory-6), and defecatory dysfunction (Colo rectal-Anal Distress Inventory-8). By adding three subscales the score ranges from 0-300. The higher the score the greater the perceived impact that pelvic floor dysfunction has on a patient's life.
Pelvic Floor Impact Questionnaire (PFQI) | Baseline to 4th Week
  The pelvic floor impact questionnaire was designed to evaluate symptoms and quality of life relating to PFDs; it included scales from the Urinary Impact Questionnaire. (UIQ-7), Pelvic Organ Prolapse Impact Questionnaire (POPIQ), Colorectal - Anal Impact Questionnaire -7(CRAIQ-7). All items use the following format with the response scale ranging from (0 to 3). Add the scores from the 3 scales together to obtain the summary score (range 0-300). Lower scores indicate less effect on QOL.
Pelvic Floor Muscle Strength Assessment through MMT-oxford scale | Baseline to 4th Week
  The grading system used to determine the strength of the pelvic floor muscles is the Oxford Scale or Modified Oxford Scale. It is a subjective grading system used to assess the strength and quality of contraction of the pelvic floor muscles. The muscles will be assessed via an external vaginal examination. Score Ranges from 0-5 . higher score indicate better muscle strength.

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Ejaz, Principal Investigator — Riphah International University
Locations (1):
- King Abdullah Teaching Hospital, Mansehra, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No